CLINICAL TRIAL: NCT05058027
Title: A Randomized, Multicenter, Subject and Assessor Blind, Parallel, Comparative Non-inferiority Clinical Trial Study to Assess the Anti-adhesive Effect and Safety of MEDICURTAIN® Applied to Undergoing Thyroid Surgery
Brief Title: Anti-adhesive Effect and Safety of MEDICURTAIN Applied to Undergoing Thyroid Surgery (Pivotal Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SPMC_0912
Record Dates: First submitted 2021-09-10; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Tissue Adhesion, Surgery-Induced
Keywords: Medicurtain®; Medicurtain; Anti-adhesion barrier; Sodium hyaluronate
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GUARDIX-SG® (Active Comparator): Treat GUARDIX-SG 6g prefilled syringe after surgery
  Interventions: Device: GUARDIX-SG®
- Medicurtain® (Experimental): Treat Medicurtain® 5ml prefilled syringe after surgery
  Interventions: Device: Medicurtain®

INTERVENTIONS:
Device: GUARDIX-SG® — GUARDIX-SG® 6g prefilled syringe
  Other Names: GUARDIX-SG
  Arms: GUARDIX-SG®
Device: Medicurtain® — Medicurtain® 5ml prefilled syringe
  Other Names: Medicurtain
  Arms: Medicurtain®

SUMMARY:
This study was designed to demonstrate the non-inferiority of MEDICURTAIN® (investigational device) compared to commercially available GUARDIX-SG® (control device) in treatment of subject who underwent total thyroidectomy for prevention of adhesion formation at 6 weeks after the surgery.

DETAILED DESCRIPTION:
This clinical trial is a randomized, multi center, subject and evaluator blinded, parallel, comparative and non-inferiority clinical trial study to assess the prevention of adhesion formation in the subjects treated either MEDICURTAIN® or GUARDIX-SG at 6 weeks after total thyroidectomy.

The primary endpoint was defined as abnormal findings of esophageal motility evaluated by the independent third evaluator using marshmallow esophagography. The objective of this study was to demonstrate the non-inferiority of investigational device versus control device for adhesion formation at 6 weeks after the administration of investigational or control devices.

Esophageal motility score and clinical symptoms assessed by the independent third evaluator using marshmallow esophagography at 6 weeks after administration of investigational device were secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. The subject (male and female) aged between 20 ~ 65.
2. The subject planned a first thyroidectomy for thyroid disease.
3. The subject did not have medical history of esophagus-related disease
4. The subject was suitable for local anesthesia or general anesthesia (Respiration and Intravenous anesthesia)
5. The subject who could communicate with the investigators fluently, understands the purpose of clinical trial and the risk of participation in the clinical trial, and was willing to comply with guideline for clinical trial.
6. The subject has been informed of the nature of the study (objective, methodology, efficacy, etc.) and signed written informed consent.
7. The subject has been informed the efficacy and risk of anesthesia related to the surgery, procedures and examination, etc. and singed written informed consent.
8. The subject who agrees to comply with permitted contraception during the study (example of permitted contraception: using condom and infertility surgery, etc.)

Exclusion Criteria:

1. The subject had general or local infection.
2. The subject was diagnosed with liver and/or kidney and coagulation abnormalities.
3. The subject took the prohibited concomitant medication.
4. The subject had suppressed immunity or autoimmune disease
5. The subject had hypersensitivity to the investigational devices.
6. The subject was pregnant of a nursing mother or those who plan pregnancy during the study.
7. The subject had serious disease that may affect to the study justified by Investigators (example: heart failure, kidney failure, pancreatitis, and diabetes, etc.)
8. The subjects participate in another investigational study after enrollment of this study or subject previously participated in another investigational study within last 3 months before participating in this study.
9. The subject considered to be not eligible to participate in the study justified by Investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-07-04 (Actual); Primary Completion 2014-08-28 (Actual); Study Completion 2014-08-28 (Actual)

PRIMARY OUTCOMES:
Presence of abnormal findings of esophageal motility evaluated by the independent third evaluator using marshmallow esophagography obtained at 6 weeks after administration of investigational device. | Week 6
  The percentage of abnormal findings measured as mild/moderate/severe in the esophageal motor performance score through marshmallow esophagography is the incidence of adhesion. The esophageal motility was scored as normal 3 point, mild 2 point, moderate 1 point and severe 0 point.

SECONDARY OUTCOMES:
Esophageal motility score assessed by the independent third evaluator using marshmallow esophagography obtained at 6 weeks after administration of investigational device | Week 6
  The esophageal motility was scored as normal 3 point, mild 2 point, moderate 1 point and severe 0 point.
Clinical Symptoms assessed using questionnaire by investigator assessed by using 10 point visual analogue scale (VAS). | Follows up to week 6
  The questionnaire is composed of three questions as shown below.
  1. Discomfort around surgical area
  2. Discomfort when a patient bends his or her neck backward
  3. Inflammation reaction and scar formation around surgical area Each item is evaluated in the 10-step evaluation of VAS. 0 = None of pain, 10 = Agonizing.
Clinical Symptoms assessed using questionnaire by subject assessed by using 10 point visual analogue scale (VAS). | Follows up to week 6
  The questionnaire is composed of four questions as shown below.
  1. Difficulty in swallowing the saliva
  2. Difficulty in swallowing the water
  3. Difficulty in swallowing the solid food
  4. Aesthetic self-satisfaction on the scar around surgical area Each item is evaluated in the 10-step evaluation of VAS. 0 = None of pain, 10 = Agonizing.

CONTACTS AND LOCATIONS:
Overall Officials: Byung In Moon, MD, PhD, Principal Investigator — Ewha Womans University Mokdong Hospital; Hang-Seok Chang, MD, PhD, Principal Investigator — Gangnam Severance Hospital; Gil Soo Son, MD, PhD, Principal Investigator — Korea University; Seung Ki Kim, MD, PhD, Principal Investigator — Cha University Bundang Cha Hospital
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, Gangnam-gu, Eonju-ro, 211, South Korea

IPD SHARING:
Plan to Share IPD: No